CLINICAL TRIAL: NCT06768229
Title: Single Arm, Open-label, Single-center Exploratory Study to Assess the Survival of Bifidobacteria's Strains in Human Gastro-intestinal Tract of Healthy Volunteers After 14 Days of Consumption of a Mix of 4 Freeze-dried Strains.
Brief Title: Survival Plant-Based
Acronym: Survi PB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23REX0060157
Record Dates: First submitted 2024-12-19; First posted 2025-01-10 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: A03 - Digestive System; B03 - Bacteria
Keywords: Strains; Survival; Bifidobacterium; Intestinal microbiota
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, single-center, exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assess the survival of Bifidobacteria's strains in the GI tract after consumption of strains mix (Experimental): One study group of 20 healthy volunteers will consume freeze-dried strains- mix twice per day diluted in 1 glass of still water during 14 consecutive days.
  Interventions: Other: Consumption of a freeze-dried strains-mix.

INTERVENTIONS:
Other: Consumption of a freeze-dried strains-mix. — One study group of 20 healthy volunteers will consume freeze-dried strains-mix twice per day diluted in 1 glass of still water during 14 consecutive days.

SUMMARY:
The aim of this study is to explore the potential of a mix of 4 freeze-dried bifidobacteria strains from Danone collection to survive in human gastro-intestinal (GI) tract of healthy volunteers after 14 days of consumption.

To this aim, one study group of 20 healthy volunteers will consume freeze-dried strains- mix twice per day diluted in 1 glass of still water during 14 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years.
2. Body Mass Index (BMI) between 18.5-30.0 kg/m2.
3. Willing to consume twice per day for at least 14 days the study product diluted in 1 glass of still water.
4. Availability to comply with the protocol and timetable.
5. Having regular bowel movements (on ≥6 days/week).
6. French speaking and reading.
7. Subject willing to adhere to the specific instructions and restrictions for the entire duration of the study.
8. Signed (written) informed consent from participant.
9. Subject is covered by a French health insurance.
10. Agree to be registered in the national database of subjects participating in clinical research.
11. Have a smartphone/computer compatible and connectable to internet, and subject is willing and able to complete the electronic Patient Reported Outcomes (ePRO) using it.
12. Women of childbearing potential must be using a medically approved method of contraception, or be with a surgically sterile partner or be with a partner of the same sex.

Exclusion Criteria:

1. Subject who used within 8 weeks prior to the screening visit or are planning to use during the conduct of this study one of the listed prohibited medications that might modify gastrointestinal function. Incidental use (1 or 2 pills/tablets) of non-steroidal anti-inflammatory drugs and aspirin is allowed, if required.
2. Subject following special diet at the screening visit (V1), or plan for such diet during the study.
3. Subject having any previous abdominal surgery, or plan for such surgery during the study.
4. Subject who underwent a general anesthesia in the preceding 4 weeks before the screening visit (V1).
5. Subject with any metabolic disease, hypertension, any inflammatory disease, any psychiatric disorder, or any gastrointestinal disorder, all these medical conditions should have been diagnosed by a physician.
6. Subject with any known food allergy or intolerance to any of the study product components or to any potential traces.
7. Active smoker with 7 or more cigarettes per week.
8. Subject doing high intensity physical activity in combination with following an enhanced diet within 1 month before screening or planned during the participation of the study.
9. Subject who underwent dental surgery within the last 4 weeks before the screening visit (V1) or plan dental surgery during the course of the study.
10. Pregnant woman or woman planning to become pregnant during the study or breastfeeding woman.
11. Participation in another study with investigational or marketed products potentially affecting the gut microbiota ≤ 4 weeks before the screening visit (V1) or plan for participation in any other intervention study during the study.
12. Employees and/or children/family members or relatives of employees of Danone Global Research & Innovation Center or the participating site.
13. Subject under guardianship or curatorship.
14. Excessive alcohol consumption during the past 6 months before the screening visit (V1).
15. Drug abuse, based on investigator's judgment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Presence of alive bacteria of each of the provided specific strains of Bifidobacterium strains in feces after 14 days of study product consumption in healthy adults. | After 14 days of study product consumption
Comparison of the quantity of total and alive bacteria of each of the provided specific strains of Bifidobacterium strains in feces before and after 14 days of study product consumption in healthy adults. | After 14 days of study product consumption
Presence of alive bacteria of the provided specific strains of each of the Bifidobacterium strains in feces after 1 week of follow-up in healthy adults. | After 1 week of follow-up
Comparison of the quantity of total and alive bacteria of each of the provided specific strains of Bifidobacterium strains in feces after 1 week of follow-up in healthy adults. | After 1 week of follow-up

SECONDARY OUTCOMES:
Dietary intakes collected by dietary recall (using MyFood24 software) of the previous day of the faecal samples collection for V2, V3 and V4 of healthy adult subjects. | After 1 week of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- CEN Experimental, Dijon, France

IPD SHARING:
Plan to Share IPD: No